CLINICAL TRIAL: NCT02488447
Title: Prospective Study for Evaluating Life Quality and Its Determinant Factors as Treatment Adherence and Immunotherapy Satisfaction in Patients With Rhinoconjunctivitis With or Without Asthma, Sensitized at Least to One Aeroallergen
Brief Title: Study for Evaluating Life Quality in Patients With Rhinoconjunctivitis
Acronym: ÍCARA
Status: Completed | Type: Observational
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: BIA-ALE-2014-01; ÍCARA (Other: Roxall Medicina España S.A.)
Record Dates: First submitted 2015-06-25; First posted 2015-07-02 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergy; Allergic rhinoconjunctivitis; Immunotherapy; Life Quality; Adherence
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of ths study is to evaluate changes in life quality of patients affected by rhinoconjuntivitis with or without asthma after immunotherapy treatment. It is an observational, prospective and comparative study before-after immunotherapy treatment with a one year follow-up.

ELIGIBILITY:
Based on Routine Clinical Practice

Inclusion criteria:

* Patients affected by allergic rhinoconjunctivitis sensityzed to one or several aeroallergens.Although allergic rhinoconjunctivitis is the pathology under study, the inclusion of patients with mild concomitant asthma is allowed (GINA 2013)
* Patients older than 12 years old
* Patients being subsidiaries of receiving allergen immunotherapy treatment
* Patients who obtained a prick test result ≥ 3 mm diameter to any aeroallergen. Positive and negative control of the test should give consistent results.
* Patients with specific immunoglobulin E ≥ class 2 (CAP/PHADIA) to any aeroallergen.

Exclusion criteria (based on routine clinical practice):

* Patients with severe asthma or forzed expiratoy volumen in 1 second FEV1< 70% even if the are pharmacologically controlled .
* Patients with: immunological, cardiac, renal or hepatic illnesses or any other medical condition that the investigator seems relevant so as to interfere with the treatment.
* Patients with a previous history of anaphylaxis
* Patients under treatment with tricyclic antidepressives, phenothiazines , β-blockers, or Angiotensin Converting Enzyme Inhibitors (ACEI)
* Female patients who are pregnant or breast-feeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by Rhinoconjunctivitis with or without asthma
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Life Quality as measured by RQLQ questionaire (≥12years) | One Year

SECONDARY OUTCOMES:
Adherence as measured by patient diary | One Year
Treatment Satisfaction as measured by visual analogue scale | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Fernández Arbeiza, Dr., Principal Investigator — Complejo Hospitalario de Cáceres; Eloína González Mancebo, Dra., Principal Investigator — Hospital Universitario de Fuenlabrada; Vanesa Sánchez, Dra., Principal Investigator — Hospital Universitario del Henares; Jose Julio Laguna, Dr., Principal Investigator — Hospital Central de la Cruz Roja; Alicia Alonso, Dra., Principal Investigator — Centro Médico Alianza Médica; Ana Mª Callejo, Dra., Principal Investigator — Hospital Virgen de la Concha; Mª Jesús Trujillo, Dra., Principal Investigator — Hospital del Tajo; Ruth Mielgo, Dra., Principal Investigator — Hospital 12 de Octubre; Javier Cuesta, Dr., Principal Investigator — Hospital Fundación Jiménez Díaz; Mónica Rodríguez, Dra., Principal Investigator — Hospital Fundación Alcorcón; Mª Antonia Padial, Dra., Principal Investigator — Hospital del Norte, Infanta Sofía; Raquel López, Dra., Principal Investigator — Complejo Hospitalario La Coruña; Carlos Colás, Dr., Principal Investigator — Hospital Clínico Lozano Blesa; Ignacio Pérez, Dr., Principal Investigator — Hospital Royo Vilanova
Locations (14):
- Spain (14):
  - Complejp Hospitalario de Cáceres, Cáceres, Extremadura
  - Complejo Hospitalario Universitario La Coruña, A Coruña, Galicia
  - Hospital Central de la Cruz Roja, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital del Tajo, Madrid
  - Hospital del Norte Infanta Sofía, Madrid
  - Hospital Universitario del Henares, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital universitario de Fuenlabrada, Madrid
  - Centro Médico Alianza Médica, Valladolid
  - Hospital Virgen de la Concha, Zamora
  - Hospital Universitario Lozano Blesa, Zaragoza
  - Hospital Royo Vilanova, Zaragoza